CLINICAL TRIAL: NCT00952224
Title: Prognostic Significance and Determinants of Myocardial Salvage Assessed by Cardiovascular Magnetic Resonance in Acute Reperfused Myocardial Infarction
Brief Title: Myocardial Salvage Assessed by Cardiovascular Magnetic Resonance - Impact on Outcome
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Other Study IDs: Leipzig MR 1
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: myocardial salvage; cardiovascular magnetic resonance; magnetic resonance imaging; myocardial infarction; prognosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute myocardial infarction patients: Patients undergoing primary percutaneous coronary intervention in ST-elevation myocardial infarction plus magnetic resonance imaging
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging — magnetic resonance imaging is used for prognosis assessment

SUMMARY:
In acute myocardial infarction cardiovascular magnetic resonance imaging can retrospectively detect the myocardium at risk and the irreversible injury. This allows for quantifying the extent of salvaged myocardium after reperfusion as a potential strong end point for clinical trials and outcome. The aim of the present study is to determine the prognostic significance and determinants of myocardial salvage assessed by CMR in reperfused ST-elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation myocardial infarction < 12 hours
* primary percutaneous coronary intervention

Exclusion Criteria:

* previous myocardial infarction
* prior fibrinolysis
* contraindications to CMR at study entry (such as implanted pacemakers, defibrillators, claustrophobia or metallic intracranial implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 6 months

SECONDARY OUTCOMES:
Mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Eitel, MD, Principal Investigator — Heart Center Leipzig - University Hospital; Holger Thiele, MD, Study Director — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] Eitel I, Desch S, de Waha S, Fuernau G, Gutberlet M, Schuler G, Thiele H. Long-term prognostic value of myocardial salvage assessed by cardiovascular magnetic resonance in acute reperfused myocardial infarction. Heart. 2011 Dec;97(24):2038-45. doi: 10.1136/heartjnl-2011-300098. Epub 2011 Oct 11. PMID 21990384
- [Derived] Eitel I, Desch S, Fuernau G, Hildebrand L, Gutberlet M, Schuler G, Thiele H. Prognostic significance and determinants of myocardial salvage assessed by cardiovascular magnetic resonance in acute reperfused myocardial infarction. J Am Coll Cardiol. 2010 Jun 1;55(22):2470-9. doi: 10.1016/j.jacc.2010.01.049. PMID 20510214